CLINICAL TRIAL: NCT03477123
Title: Evaluation of Robotic Exoskeletons Therapy for Gait Rehabilitation in Patients With Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nacional de Parapléjicos de Toledo (Other)
Collaborators: Institut Guttmann (Other)
Responsible Party: Principal Investigator, Angel Gil-Agudo, PhD, MD, Head of Rehabilitation, Hospital Nacional de Parapléjicos de Toledo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/01437
Record Dates: First submitted 2018-02-28; First posted 2018-03-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Spinal Cord Injury; Incomplete Spinal Cord Injury
Keywords: Incomplete spinal cord injury; Walking; Rehabilitation; Robotic exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator does not have information on the group the patient was enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Walking therapy with Exo-H2 exoskeleton
  Interventions: Device: Walking therapy with Exo-H2 exoskeleton
- Control (No Intervention): Group receiving conventional walking therapy without robotic exoskeleton

INTERVENTIONS:
Device: Walking therapy with Exo-H2 exoskeleton
  Arms: Intervention

SUMMARY:
The objective of the study is to assess the efficacy of the Exo-H2 robotic exoskeleton for walking rehabilitation of people with incomplete spinal cord injury.

DETAILED DESCRIPTION:
The recovery of walking ability is a primary concern of rehabilitation programs for people who have suffered anincomplete spinal cord injury. Robotic therapy arises from the new concepts of neuroplasticity. One of the most novel contributions in this field is robotic exoskeletons. However, there is still not enough scientific evidence to support the clinical use of this technology.

The aim of this proposal is to assess the efficacy of a new model of robotic exoskeleton (Exo H2) developed by the CSIC with HNP involvement in the context of HYPER project (Consolider 2009 call) in gait rehabilitation for people with incomplete spinal cord injury. A multicenter study is proposed here, involving the National Hospital of Paraplegics and the Institut Guttmann. Two randomized groups of patients with subacute incomplete spinal cord injury will be defined. In one group, protocol gait rehabilitation based on the Exo H2 will be established and traditional gait therapy will be adapted for control group. Both groups of patients were assessed performing a physical exam including functional gait scales (10 MWT, 6MWT, WISCI II score, SCIM) and a biomechanical gait analysis with kinetic and kinematic techniques. Functional assessment will be carried out before intervention, at the end of the intervention and a follow up six weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete Spinal Cord Syndrome, ASIA scale C or D
* enough strength in the upper extremities to handle a walker or crutches (triceps brachial muscle balance ≥ 3)
* Age between 16 and 70 y.o.
* Heigth: 1.6-1.9m
* Weigth less than 120Kg
* Stable medical condition between 6 weeks and 18 months since injury.
* Subjects must tolerate standing and be included in walking rehabilitation program in the center.
* Lower limb spasticity should be lower than 3 as measyred by Ashworth scale.

Exclusion Criteria:

* Cardiovascular diseases.
* Upper limb pathology of any kind.
* irreducible flexo or arthrodesis in lower limb joints, 2 or more osteoporotic fractures in the lower limbs in the last 2 years
* Uncontrolled epilepsy.
* Ulcers sores at the contact points with the exoskeleton.
* Refuse to participate.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Lower extremity motor score | Change from Baseline Lower Extremity Motor Score at 2 months
  This scale evaluate the ability and force of the patient when attepmting to contract five key lower limb muscles. It is manually measured by the therapist. Range from 0 (no contraction) to 5 (healthy function). The total score summs up the scores of all muscles. In healthy conditions is 50 points.
Spasticity measured by Ashworth scale | Change from Baseline Ashworth Scale at 2 months
  Manual testing of muscle tone in response to manual mobilization of joints. Range from 0 (healthy response) to 4 (maximum muscle tone).
Ten meters walking test | Change from Baseline Ten Meters Walking Test at 2 months
  This test measure walking velocity on covering ten meters walking in flat, straigth line.
Six minutes walking test | Change from Baseline Six Minutes Walking Test at 2 months
  This test measure walking endurance by measuring the distance covered in six minutes of walking in flat, straigth line.
Time Up-and-Go Test (TUG) | Change from Baseline TUG Test at 2 months
  This test measures the time to complete stand to sit, walk 3 meters and sitting back again.
Walking Index for Spinal Cord Injury II (WISCI II) | Change from Baseline WISCI II Scale at 2 months
  WISCI II assess the amount of physical assistance needed, as well as devices required, for walking following paralysis that results from Spinal Cord Injury.
  The subject is observed by the trained personnel and the WISCI level is recorded on the scale of 0 to 20 at baseline (Baseline WISCI). The subject is observed again at the defined interval (Interval WISCI). The change in score is calculated by subtracting the baseline WISCI from the Interval WISCI, which equals the change in WISCI (Changed WISCI). If a group of subjects are enrolled, medians and means may be calculated.
Questionnaire: Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Through study completion
  The purpose of the QUEST questionnaire is to evaluate how satisfied you are with your assistive device and the related services you experienced. The questionnaire consists of 12 satisfaction items. For each of the 12 items, rate your satisfaction with your assistive device and the related services you experienced by using the following scale of 1 to 5.

SECONDARY OUTCOMES:
Spinal Cord Independence Measure III (SCIM III) | Change from Baseline SCIM III scale at 2 months
  The SCIM is composed of 19 items that assess 3 domains.1) Self-care, 2) Respiration and sphincter management, 3) Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Gil-Agudo, PhD, MD, Study Chair — Head of Rehabilitation Department
Locations (1):
- National Hospital for Paraplegics, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ditunno PL, Patrick M, Stineman M, Ditunno JF. Who wants to walk? Preferences for recovery after SCI: a longitudinal and cross-sectional study. Spinal Cord. 2008 Jul;46(7):500-6. doi: 10.1038/sj.sc.3102172. Epub 2008 Jan 22. PMID 18209742
- [Background] Esquenazi A, Packel A. Robotic-assisted gait training and restoration. Am J Phys Med Rehabil. 2012 Nov;91(11 Suppl 3):S217-27; quiz S228-31. doi: 10.1097/PHM.0b013e31826bce18. PMID 23080038
- [Background] Kwakkel G, Kollen B, Lindeman E. Understanding the pattern of functional recovery after stroke: facts and theories. Restor Neurol Neurosci. 2004;22(3-5):281-99. PMID 15502272
- [Background] Chen G, Patten C. Treadmill training with harness support: selection of parameters for individuals with poststroke hemiparesis. J Rehabil Res Dev. 2006 Jul-Aug;43(4):485-98. doi: 10.1682/jrrd.2005.04.0063. PMID 17123188
- [Background] Colombo G, Joerg M, Schreier R, Dietz V. Treadmill training of paraplegic patients using a robotic orthosis. J Rehabil Res Dev. 2000 Nov-Dec;37(6):693-700. PMID 11321005
- [Background] Mantone J. Getting a leg up? Rehab patients get an assist from devices such as HealthSouth's AutoAmbulator, but the robots' clinical benefits are still in doubt. Mod Healthc. 2006 Feb 13;36(7):58-60. No abstract available. PMID 16515076
- [Background] Veneman JF, Kruidhof R, Hekman EE, Ekkelenkamp R, Van Asseldonk EH, van der Kooij H. Design and evaluation of the LOPES exoskeleton robot for interactive gait rehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2007 Sep;15(3):379-86. doi: 10.1109/tnsre.2007.903919. PMID 17894270
- [Background] Tefertiller C, Pharo B, Evans N, Winchester P. Efficacy of rehabilitation robotics for walking training in neurological disorders: a review. J Rehabil Res Dev. 2011;48(4):387-416. doi: 10.1682/jrrd.2010.04.0055. PMID 21674390
- [Background] Zeilig G, Weingarden H, Zwecker M, Dudkiewicz I, Bloch A, Esquenazi A. Safety and tolerance of the ReWalk exoskeleton suit for ambulation by people with complete spinal cord injury: a pilot study. J Spinal Cord Med. 2012 Mar;35(2):96-101. doi: 10.1179/2045772312Y.0000000003. Epub 2012 Feb 7. PMID 22333043
- [Background] Aach M, Cruciger O, Sczesny-Kaiser M, Hoffken O, Meindl RCh, Tegenthoff M, Schwenkreis P, Sankai Y, Schildhauer TA. Voluntary driven exoskeleton as a new tool for rehabilitation in chronic spinal cord injury: a pilot study. Spine J. 2014 Dec 1;14(12):2847-53. doi: 10.1016/j.spinee.2014.03.042. Epub 2014 Apr 4. PMID 24704677
- [Background] Jackson AB, Carnel CT, Ditunno JF, Read MS, Boninger ML, Schmeler MR, Williams SR, Donovan WH; Gait and Ambulation Subcommittee. Outcome measures for gait and ambulation in the spinal cord injury population. J Spinal Cord Med. 2008;31(5):487-99. doi: 10.1080/10790268.2008.11753644. PMID 19086706
- [Background] Ditunno J, Scivoletto G. Clinical relevance of gait research applied to clinical trials in spinal cord injury. Brain Res Bull. 2009 Jan 15;78(1):35-42. doi: 10.1016/j.brainresbull.2008.09.003. Epub 2008 Oct 9. PMID 18848865